CLINICAL TRIAL: NCT00525980
Title: Interactive CD-ROM on Cancer Genetics for Hispanics
Brief Title: Cancer Genetics CD-ROM for Hispanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0339
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Cancer Risk; CD-ROM; Focus Group; Cancer Genetics
MeSH Terms: conditions — Breast Neoplasms | interventions — Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: Written Materials (Experimental): One group asked to read educational materials.
  Interventions: Behavioral: Focus Group; Other: Written Materials; Behavioral: Questionnaires
- Group 2: Computer Program Only (Experimental): Group 2 use an educational computer program to learn about breast cancer risk and genetic testing without guidance.
  Interventions: Behavioral: Computer Program; Behavioral: Focus Group; Behavioral: Questionnaires
- Group 3: Computer Program + Promotora (Experimental): Group 3 use the computer program with the guidance of a promotora.
  Interventions: Behavioral: Computer Program; Behavioral: Focus Group; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Computer Program — Participants will be given a program to learn about breast cancer risk and genetic testing.
  Arm 3 Only = Participants will use the program with the assistance of a promotora (female "promoter," community health worker, sometimes known as a lay health advisor).
  Arms: Group 2: Computer Program Only; Group 3: Computer Program + Promotora
Behavioral: Focus Group — Focus group discussion lasting about 60 to 90 minutes.
Other: Written Materials — Printed materials will be given. The CD-ROM will be offered at the end of the study.
  Arms: Group 1: Written Materials
Behavioral: Questionnaires — Occasional questionnaire, written or verbal phone survey, about knowledge and attitudes toward cancer and genetic testing.
  Other Names: Survey

SUMMARY:
This project will build upon prior, successful research on the effectiveness of an interactive computer disk with readable only memory (CD-ROM) for educating women about breast cancer and genetic risk. Prior studies found that an interactive CD-ROM for educating women about breast cancer risk and genetic testing was effective. The program was well received by lay persons and professionals. In a randomized controlled trial conducted at multiple sites, the CD-ROM intervention was highly effective in increasing knowledge, especially among women at low risk of carrying a breast cancer susceptibility gene 1/2 (BRCA1/2) mutation.

Researchers now propose to expand the use of the interactive CD-ROM in two innovative ways. The overall goal of this proposal is to evaluate the program as a first-line educational approach for Hispanic women on the Texas-Mexico border, where educational resources about cancer genetics are limited. First, researchers will modify and adapt the program for a primarily Hispanic population, in order to make it culturally and linguistically appropriate to the needs of that audience.

Second, researchers will evaluate the program as a first-line educational method among women with a personal or family history of breast cancer. Researchers will compare the effectiveness of the CD-ROM when implemented with and without the guidance of a trained promotora, and in comparison with standard educational materials (usual care condition).

The specific aims of this study include:

Aim 1: To modify the interactive CD-ROM to: a) make it culturally and linguistically appropriate for Hispanic women residing along the Texas-Mexico border; b) reflect current knowledge about breast cancer genetics; c) add a module to help women prepare to discuss their family history and cancer risk with a health care provider (n=50 participants).

Aim 2: To conduct a randomized, controlled evaluation that compares the efficacy of the modified CD-ROM when used alone vs. when used with a promotora-assisted approach vs. standard written materials (n=414 participants).

DETAILED DESCRIPTION:
This study will test ways to help improve Hispanic women's knowledge and understanding about breast cancer risk and genetic testing for inherited cancer risk. These methods include providing printed educational materials, using an educational computer program, and using the computer program with the assistance of a lay health worker (a promotora).

If you agree to take part in this study, you will complete a questionnaire that will ask about your personal health as well as your knowledge and attitudes toward cancer and genetic testing. After the questionnaire is completed, you will be randomly assigned (as in the roll of dice) to 1 of 3 study groups. One group will be asked to read educational materials. Another group will use an educational computer program to learn about breast cancer risk and genetic testing without guidance. Another group will use the computer program with the guidance of a promotora.

Each of the 3 study groups should take between 30 and 60 minutes to complete.

Immediately after participating in your assigned group, you will be asked to complete another questionnaire that will ask about your knowledge and attitudes toward cancer and genetic testing. You will also be contacted later by telephone to complete similar questionnaires at about 1 month and 6 months after your study visit. Some women will be asked to complete an additional questionnaire by telephone 1 week after reading the educational materials or the computer program, and researchers will ask for permission to audiotape this interview. It will take about 20 minutes to complete each of the questionnaires used in this study.

This is an investigational study. Up to 414 women will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* Residing in the El Paso metropolitan area and self-identifying as Hispanic
* Being 18 years of age or older
* Women who have a personal history of breast cancer or have a first-degree relative with breast cancer OR lay health workers (male or female)
* Able to provide informed consent

Exclusion Criteria:

* Having a primary language other than English or Spanish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Data analysis of structured questionnaires | 3 Years

SECONDARY OUTCOMES:
Comparison of 3 Intervention Groups by Continuous Outcomes (knowledge, risk assessment, decisional conflict and quality of life) | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Peterson, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - The Cancer and Chronic Disease Consortium (CCDC) of El Paso, El Paso, Texas
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org